CLINICAL TRIAL: NCT04747210
Title: Improving Students' Participation in Daily Living Skills Through Contextual Coaching One-on-one for Special Needs Assistants.
Brief Title: Contextual Coaching Versus Training Workshop for Assistants in Special Education.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Maria Jose López-de-la-Fuente, Occupational Therapist. Departamento de Fisiatría y Enfermería, Universidad de Zaragoza
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COACHvsW
Record Dates: First submitted 2021-01-30; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Disabled Persons; Caregiver
Keywords: Special Need Assistants/paraprofessionals; Coaching; Occupational therapy; Self-care skills

STUDY DESIGN:
Intervention Model Description: This study is a quasi-experimental pretest-posttest design. Repeated measures on participants in both arms (as in an RCT) enable assessment of both within-person changes over time and between-arm differences.
Who Masked: Outcomes Assessor
Masking Description: Two external assessors will measure the fidelity of the implementation of the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trainig workshop and Coaching one-on-one (Active Comparator): Ten-hour training workshop that was divided into three sessions outside working hours. Coaching one-on-one in the daily routines and natural environment.
  Interventions: Behavioral: contextual one-on-one coaching
- Trainig workshop (Active Comparator): Assistants receive ten-hour training workshop that was divided into three sessions outside working hours.
  Interventions: Behavioral: Trainig workshop

INTERVENTIONS:
Behavioral: contextual one-on-one coaching — Training workshop and coaching one-on-one
  Arms: Trainig workshop and Coaching one-on-one
Behavioral: Trainig workshop — Ten-hour training workshop.
  Arms: Trainig workshop

SUMMARY:
Special Need Assistants/paraprofessionals serve an essential role in special education to support children with multiple disabilities, but they often lack adequate training and supervision. The study aims to examine the effects of the coaching program for assistants compared to a workshop outside working hours and evaluate the outcomes in students and assistants. The second aim is to measure fidelity implementation of coaching practices and if the intervention was participation-based.

DETAILED DESCRIPTION:
This study addresses the training needs of assistants to minimize participation barriers of the students. The schools will be assigned to one of two groups: both groups will receive a 10 hours training workshop; only the intervention group will receive coaching one-to-one. The duration and number of coaching sessions will depend on the caregivers' time available, daily routines, and goals. Coaching sessions will be recorded for the assessment of treatment fidelity.

ELIGIBILITY:
Inclusion Criteria assistants:

* Special Need Assistant of students between 4-21 years of age.
* Speak, read and comprehend Spanish.
* Be available for workshop and one-on-one coaching.
* Able to verbalize changes in their own performance or their students' participation.
* Written consent.

Exclusion Criteria assistants:

* Have no students involved in the program.

Inclusion Criteria students:

* Present difficulties in Activities of Daily Living (ADLs).
* Have an assistant involved in the study.
* Informed consent signature (parents or legal tutors).

Exclusion Criteria students:

* Independence in activities of daily living.
* 70 or more points in the Care Dependency Scale for Pediatrics (CDS-P).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Change in The Canadian Occupational Performance Measure (COPM). Students | baseline- 3 month after intervention
  Caregivers identify activities that are problematic for the child. The caregiver rates the child's performance and satisfaction for each participation goal on a 10-point scale, (1=unable to perform, unsatisfied; 10= performs exceptionally well, extremely satisfied). Differences in scores pre-and post-intervention for both performance and satisfaction are determined independently. A 2-points change in these values is considered clinically meaningful.
Change in Goal Attainment Scaling (GAS). Assistants. | Baseline - 3 month after intervention
  Clients identify goals and rate their performance on a 5-point Likert scale ranging from -2 (much less than expected) to +2 (much better than expected). In the baseline, clients can score -1 or -2, and the score "0" is the expected level of success. The 4-point Likert scale is used for quantifying importance (ranging from 0= nothing important to 3= really important) and difficulty (ranging from 0= easy to 3= very difficult). Afterwards, the goal's weight is calculated (importance*difficulty). A mathematical formula allows computation to T-score with a mean of 50 and a standard deviation of 10.

SECONDARY OUTCOMES:
The Coaching Practices Rating Scale. | 12 month after intervention
  The Coaching Practices Rating Scale was utilized as a secondary outcome to measure the fidelity of coaching. Its 14 items are based on adults' learning characteristics and coaching practices to determine how the coach use these practices, on a 5-point Likert scale. The scale accepts the rating through video-tapes and has a high degree of construct validity and internal consistency.
Natural Environments Rating Scale (NERS) | 12 month after intervention
  The NERS describes eight categories: 1) setting; 2) activity; 3) type of activity; 4) engagement of child; 5) activity leader; 6) materials; 7) role of the caregiver; 8) the role of the professional. If there is no child-centred activity, grading is discontinued for the remaining categories. Only the last four categories are rated for an overall score that differentiated traditional or participation-based services.
Change in learning. Social validity | 6 month
  Paraprofessionals were invited to reply to a writing questionnaire. This survey collected information about their training preferences and satisfaction with received training.
Change in transfer and generalization of learning | 19-20 mounths after intervention
  All paraprofessionals were invited to reply to a semi-structured interview through a phone. This interview collected information about their current employment, the degree in which they had been able to put into practice the skills learned and the challenges for their professional development.

OTHER OUTCOMES:
Classification of goals and adaptations | 6 month
  The types of goals and adaptations were classified according to daily living activities, such as using the toileting, eating, feeding, hygiene and grooming, dressing, functional mobility, and others (miscellanea). Accommodations or adaptations to enhance children's participation were registered during and after the intervention as a) not necessary, b) natural for the child or easy to acquire, c) a rehabilitation device, or d) an architectonic/extensive modification. The adaptations were analyzed as an independent element in the goals that improved performance two or more points in the COPM.

CONTACTS AND LOCATIONS:
Overall Officials: Maria J López-de-la-Fuente, Principal Investigator — Departamento de Fisiatría y Enfermería. Universidad de Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez-de-la-Fuente MJ, Herrero P, Garcia-Foncillas R, Gomez-Trullen EM. Contextual, Client-Centred Coaching Following a Workshop: Assistants Capacity Building in Special Education. Int J Environ Res Public Health. 2021 Jun 11;18(12):6332. doi: 10.3390/ijerph18126332. PMID 34208053